CLINICAL TRIAL: NCT06792695
Title: A Phase II, Open-label, Multicenter, Master Protocol to Evaluate the Safety and Efficacy of Novel Study Interventions and Combinations in Participants With Colorectal Cancer (CANTOR)
Brief Title: A Study of Novel Study Interventions and Combinations in Participants With Colorectal Cancer
Acronym: CANTOR
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D798VC00001; 2024-518469-84 (Registry Identifier: EU (CTIS))
Record Dates: First submitted 2025-01-20; First posted 2025-01-27 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Metastatic disease; Immunotherapy; Liver metastasis; Mismatch-repair-proficient; Antibody targeting; Colorectal Cancer; CANTOR
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — Fluorouracil; Leucovorin; Irinotecan; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Volrustomig + FOLFIRI+ Bevacizumab group (Arm A) (Experimental): Participants will receive FOLFIRI and bevacizumab together with volrustomig.
  Interventions: Drug: Volrustomig; Drug: FOLFIRI (Fluorouracil (5-FU), leucovorin, irinotecan); Drug: Bevacizumab
- FOLFIRI+ BEVACIZUMAB group (Arm B) (Active Comparator): Partcipants will receive FOLFIRI and bevacizumab.
  Interventions: Drug: FOLFIRI (Fluorouracil (5-FU), leucovorin, irinotecan); Drug: Bevacizumab

INTERVENTIONS:
Drug: Volrustomig — Volrustomig will be administered as intravenous (IV) infusion.
  Other Names: MEDI5752
  Arms: Volrustomig + FOLFIRI+ Bevacizumab group (Arm A)
Drug: FOLFIRI (Fluorouracil (5-FU), leucovorin, irinotecan) — FOLFIRI will be administered as IV infusion.
Drug: Bevacizumab — Bevacizumab will be administered as IV infusion.

SUMMARY:
The main purpose of this study is to evaluate the safety and efficacy of novel study interventions and combinations in participants with Colorectal Cancer (CRC).

DETAILED DESCRIPTION:
This is a Phase II, platform, open-label, multi-drug, multicenter, global study.

This is a modular study, that includes a master protocol and substudies.

Partcipants will be randomised to one of the following intervention groups:

* Volrustomig + FOLFIRI + bevacizumab group (Arm A)
* FOLFIRI + bevacizumab group (Arm B)

The substudy will evaluate the effects of volrustomig in combination with FOLFIRI (irinotecan, 5-FU, and leucovorin) and bevacizumab versus FOLFIRI and bevacizumab only in participants with Mismatch-repair-proficient (pMMR)/Microsatellite stable (MSS) metastatic CRC (mCRC) in the absence of liver metastases and who have not received previous systemic treatment for advanced or metastatic disease.

ELIGIBILITY:
Overall Inclusion Criteria:

* Histopathologically confirmed colorectal adenocarcinoma.
* Provision of FFPE tumor sample collected as per SoC.
* Presence of measurable disease by RECIST 1.1 criteria.
* ECOG performance status of 0 or 1.
* Life expectancy ≥ 12 weeks at the time of screening.

Substudy Inclusion Criteria:

* No radiological evidence of liver metastasis.
* No prior systemic therapy for mCRC, except for neoadjuvant/adjuvant chemotherapy where, > 6 months have elapsed between completion of therapy and documented date of diagnosis of recurrent or metastatic disease.
* Known pMMR/MSS status (only pMMR/MSS mCRC allowed).
* Adequate organ and bone marrow function
* Body weight > 35 kg at screening and at randomization.
* Contraceptive use by participants should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

Overall Exclusion Criteria:

* Central nervous system metastases or spinal cord compression
* Known history of severe allergy to any monoclonal antibody or study intervention.
* Any unresolved toxicity CTCAE Grade ≥ 2 from a previous anticancer therapy.
* History of another primary malignancy.

Substudy Exclusion Criteria:

* Potentially resectable disease with multidisciplinary plan for radical surgery.
* Active or prior documented autoimmune or inflammatory disorders or cardiac conditions.
* Participants with a prior history of hypertensive crisis or hypertensive encephalopathy or bleeding risks.
* Deep venous thrombosis, pulmonary embolism, arterial thrombosis, transient ischemic attack or cerebrovascular accident.
* History of abdominal or tracheoesophageal fistula, GI perforation and/or fistulae, or intraabdominal abscess within 6 months prior to randomization.
* Prior exposure to immune mediated therapy.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-03-12 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2028-06-07 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Approximately 3 years
  PFS is defined as the time from randomization until progression per Response Evaluation Criteria in Solid Tumours, Version 1.1 (RECIST 1.1) or death due to any cause.
Number of Participants with Adverse Events (AEs) | Approximately 3 years
  Number of participants who received at least one dose of study treatment will be assessed.

SECONDARY OUTCOMES:
Overall Survival (OS) | Approximately 3 years
  OS is defined as the time from randomization until the date of death due to any cause.
Objective Response Rate (ORR) | Approximately 3 years
  ORR is defined as the proportion of participants who have a confirmed complete response or confirmed partial response as per RECIST 1.1.
Disease Control Rate (DCR) | Approximately 3 years
  DCR is defined as the percentage of participants who have a confirmed CR or PR or who have SD per RECIST 1.1 after randomization.
Duration of Response (DOR) | Approximately 3 years
  DoR is defined as the time from the date of first documented confirmed response until date of documented progression per RECIST 1.1 or death due to any cause.
Time to second progression or death (PFS2) | Approximately 3 years
  PFS2 is defined as the time from randomization to the earliest of the progression event, after first subsequent therapy, or death.
Maximum Observed Concentration (Cmax) | Approximately 3 years
  Concentration of novel study intervention in serum and PK parameters as data allow (such as peak and trough concentrations) will be assessed.
Observed lowest concentration before the next dose is administered (Ctrough) | Approximately 3 years
  Concentration of novel study intervention in serum and PK parameters as data allow (such as peak and trough concentrations) will be assessed.
Number of patients with positive Antidrug Antibodies (ADAs) | Approximately 3 years
  The immunogenicity (ADAs) of novel study intervention in participants with CRC in the absence of liver metastases is investigated.

CONTACTS AND LOCATIONS:
Locations (65):
- United States (14):
  - Research Site, Scottsdale, Arizona
  - Research Site, Los Angeles, California
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Chicago, Illinois
  - Research Site, Baltimore, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Rochester, Minnesota
  - Research Site, Trenton, New Jersey
  - Research Site, Rochester, New York
  - Research Site, Cleveland, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Nashville, Tennessee
  - Research Site, Houston, Texas
- Australia (3):
  - Research Site, East Melbourne
  - Research Site, Wollongong
  - Research Site, Woodville South
- Canada (4):
  - Research Site, Victoria, British Columbia
  - Research Site, Barrie, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
- China (6):
  - Research Site, Beijing
  - Research Site, Chengdu
  - Research Site, Harbin
  - Research Site, Shanghai
  - Research Site, Wuhan
  - Research Site, Zhengzhou
- France (6):
  - Research Site, Bordeaux
  - Research Site, Marseille
  - Research Site, Montpellier
  - Research Site, Poitiers
  - Research Site, Saint-Priez En Jarez
  - Research Site, Villejuif
- Germany (5):
  - Research Site, Berlin
  - Research Site, Dresden
  - Research Site, Essen
  - Research Site, Hamburg
  - Research Site, Marburg
- Italy (8):
  - Research Site, Bologna
  - Research Site, Castelfranco Veneto
  - Research Site, Florence
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Pavia
  - Research Site, Pisa
  - Research Site, Roma
- Netherlands (3):
  - Research Site, Amsterdam
  - Research Site, Maastricht
  - Research Site, Zwolle
- South Korea (2):
  - Research Site, Seoul
  - Research Site, Yongin-si
- Spain (6):
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Pamplona
  - Research Site, Santander
  - Research Site, Valencia
- Taiwan (4):
  - Research Site, Kaohsiung City
  - Research Site, Taipei
  - Research Site, Taoyuan District
  - Research Site, Yung Kang City
- United Kingdom (4):
  - Research Site, Cambridge
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Metropolitan Borough of Wirral

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes",indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure researchenvironmentVivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/